CLINICAL TRIAL: NCT04408105
Title: Study of Compliance, Practice Patterns, and Barriers REgarding Established National Screening Programs for Barrett's Esophagus: SCREEN-BE
Brief Title: Survey Study on Barrett's Esophagus Screening
Acronym: SCREEN-BE
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: American College of Gastroenterology (Other)
Responsible Party: Sponsor
Other Study IDs: 19-3052.cc; NCI-2020-13912 (Other: CTRP)
Record Dates: First submitted 2020-05-11; First posted 2020-05-29 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Gastroesophageal Reflux Disease; Barrett's Esophagus; Esophagus Adenocarcinoma
Keywords: Barrett's Esophagus; Upper Endoscopy; Barrett's Esophagus Screening; GERD; Gastroesophageal Reflux Disease; BE; EAC; Esophageal Adenocarcinoma
MeSH Terms: conditions — Gastroesophageal Reflux; Barrett Esophagus; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Primary Care Providers: 400 eligible primary care providers (PCPs) will be recruited across the 7 participating sites to complete an anonymous survey. The survey will be distributed to eligible PCPs by the study site research coordinator via anonymous REDCap internet survey with 2 additional automated electronic reminders. There will also be opportunities for providers to complete a paper survey at PCP clinic meetings which will be collected by only the site research coordinator to maintain response anonymity.
  Interventions: Behavioral: Primary Care Provider Survey
- Gastroenterologists: 100 eligible gastroenterologists (GIs) will be recruited across the 7 participating sites to complete an anonymous survey. The survey will be distributed to eligible GIs by the study site research coordinator via anonymous REDCap internet survey with 2 additional automated electronic reminders. There will also be opportunities for GIs to complete a paper survey at provider clinic meetings which will be collected by only the site research coordinator to maintain response anonymity.
  Interventions: Behavioral: Gastroenterologist Survey
- Patients: 500 eligible patients will be recruited across the 7 participating sites to complete a survey. The survey will be distributed to eligible patients at the time of a clinic appointment, via telephone, or via a REDCap internet survey that will allow for 2 additional electronic phone call reminders and 1 email reminder.
  Interventions: Behavioral: Patient Survey

INTERVENTIONS:
Behavioral: Primary Care Provider Survey — To assess PCP demographics, attitudes, and perceived barriers to BE screening, we have developed a PCP survey using a theoretical model of physician behavior based on Social Cognitive Theory and the Theory of Reasoned Action. This approach has proven effective in colorectal cancer and hepatocellular carcinoma screening. This model includes domains of provider background and experience, screening practices, perceptions of screening, physician influences, and practice environment and practice patterns. To assess PCP knowledge of BE screening, we have designed 9 clinical vignettes that will categorize provider responses into under-, appropriate, and over-use of BE screening. Survey questions and vignettes have been adapted from earlier validated surveys. Prior to distribution, the survey and vignettes will be pretested and refined based on a cognitive interview about the survey among a convenience sample of 10 PCPs.
  Groups: Primary Care Providers
Behavioral: Gastroenterologist Survey — To assess GI demographics, attitudes, and perceived barriers to BE screening, we have developed a GI survey using a theoretical model of physician behavior based on Social Cognitive Theory and the Theory of Reasoned Action. This approach has proven effective in colorectal cancer and hepatocellular carcinoma screening. This model includes domains of provider background and experience, screening practices, perceptions of screening, physician influences, and practice environment and practice patterns. To assess GI knowledge of BE screening, we have designed 9 clinical vignettes that will categorize provider responses into under-, appropriate, and over-use of BE screening. Survey questions and vignettes have been adapted from earlier validated surveys. Prior to distribution, the survey and vignettes will be pretested and refined based on a cognitive interview about the survey among a convenience sample of 10 GIs.
  Groups: Gastroenterologists
Behavioral: Patient Survey — To assess patient knowledge, attitudes, and barriers to completion of BE screening, we will use a theoretical model of patient behavior on the Health Behavior Framework to guide selection of relevant variables for survey development including 4 domains: knowledge about BE and EAC, potential barriers to BE screening completion, patient attitudes and demographic information. Prior to distribution, the survey will be refined and pretested among a sample of 10 patients with each participant completing a cognitive interview prior to distribution.
  Groups: Patients

SUMMARY:
The goal of this study is to optimize Barrett's Esophagus (BE) screening to reduce the incidence, morbidity, and mortality of Esophageal Adenocarcinoma (EAC).

DETAILED DESCRIPTION:
The initial step to achieve this goal is to study shortcomings of the current BE screening referral processes in the United States. These shortcomings will be identified through completion of two synergistic aims that assess:, (1) provider knowledge, attitudes, and barriers to BE screening referral and (2) patient knowledge, attitudes, and barriers to completion of BE screening. The central hypothesis is that there are patient- and provider-level factors that can be modified to improve BE screening adherence. This hypothesis was formulated based on strong preliminary data demonstrating significant single-mindedness among gastroenterologists regarding BE screening criteria.

ELIGIBILITY:
1. Patient Eligibility Criteria

   Inclusion Criteria:
   * Patients identified by ICD-10 codes for GERD (K21.0 and K21.9) AND
   * Have had at least one outpatient clinic visit at a participating site

   Exclusion Criteria:
   * Prior diagnosis of BE/EAC
   * Non-English speaking
2. Provider Eligibility Criteria

Inclusion Criteria:

* Provider must be a PCP and/or gastroenterologist AND
* Must be at a participating site

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. We will include patients with a diagnosis of gastroesophageal reflux disease (GERD) who have at least one outpatient clinic visit at a participating site. Patients will be identified through an administrative query of the electronic medical record by ICD-10 codes for GERD (K21.0 and K21.9) as well as through a review of the upcoming clinic schedule. Patients with prior diagnosis of BE/EAC or language other than English will be excluded. Across the 7 sites, we plan to enroll 500 patients.
  2. This study will include PCPs and gastroenterologists at participating sites. Across the 7 participating centers, we plan to enroll 100 gastroenterologists and 400 PCPs.
Sampling Method: Non-Probability Sample
Enrollment: 725 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
To define provider-level knowledge, attitudes, and barriers to BE screening. | 2 years
  This investigator will conduct a survey study among primary care providers and gastroenterologists at 7 large health systems in the U.S.-including 4 tertiary care referral centers and 3 safety-net health systems. Based on constructs from Social Cognitive Theory and Theory of Reasoned Action, the survey will assess provider knowledge, attitudes, and barriers to BE screening among at-risk individuals.
To characterize the association between patient-level knowledge, attitudes, and barriers regarding BE screening. | 2 years
  This investigator will conduct a survey study among patients at 7 large health systems in the U.S. Based on constructs from the Health Behavior Framework, the survey will assess patient knowledge, attitudes, and barriers to BE screening. To accomplish these study aims, this investigator has assembled a strong and diverse team with complementary areas of expertise in Barrett's esophagus, and survey research.

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Wani, MD, Principal Investigator — University of Colorado, Denver
Locations (7):
- United States (7):
  - Denver Health Medical Center, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Pennsylvania Presbyterian Hospital, Philadelphia, Pennsylvania
  - Parkland Health and Hospital System, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kolb JM, Chen M, Tavakkoli A, Gallegos J, O'Hara J, Tarter W, Hochheimer CJ, Golubski B, Kopplin N, Hennessey L, Kalluri A, Devireddy S, Scott FI, Falk GW, Singal AG, Vajravelu RK, Wani S. Patient Knowledge, Risk Perception, and Barriers to Barrett's Esophagus Screening. Am J Gastroenterol. 2023 Apr 1;118(4):615-626. doi: 10.14309/ajg.0000000000002054. Epub 2022 Oct 11. PMID 36219171